CLINICAL TRIAL: NCT05147701
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cells for the Treatment of Non-arteritic Ischemic Optic Neuropathy
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cells for NAION
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-1-MSC-014
Record Dates: First submitted 2021-11-29; First posted 2021-12-07 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Eye Diseases; Retinitis Pigmentosa; Diabetic Retinopathy; Macular Degeneration; Traumatic Optic Neuropathy; Optic Atrophy
Keywords: Eye Diseases; Retinitis Pigmentosa; stem cell treatment; Diabetic Retinopathy; Macular Degeneration; Traumatic Optic Neuropathy; Optic Atrophy
MeSH Terms: conditions — Eye Diseases; Retinitis Pigmentosa; Diabetic Retinopathy; Macular Degeneration; Optic Nerve Injuries; Optic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (AlloRx) (Experimental): intravenous and sub-tenon delivery (total dose of 100 million cells)
  Interventions: Biological: AlloRx

INTERVENTIONS:
Biological: AlloRx — cultured allogeneic adult umbilical cord derived mesenchymal stem cells

SUMMARY:
This trial will study the safety and efficacy of intravenous and sub-tenon delivery of cultured allogeneic adult umbilical cord derived mesenchymal stem cells for the treatment of non-arteritic ischemic optic neuropathy

DETAILED DESCRIPTION:
This patient funded trial aims to study the safety and efficacy of intravenous and sub-tenon delivery of cultured allogeneic adult umbilical cord derived mesenchymal stem cells (UC-MSCs) for the treatment of non-arteritic ischemic optic neuropathy. The total dose will be 100 million cells. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

For patients with more severe disease an autologous Effector cells (activated lymphocytes) treatment will be utilized created from the patient's own cells obtained by apheresis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of NAION (non-arteritic ischemic optic neuropathy)
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (2):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Center for Investigation in Tissue Engineering and Cellular Therapy, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung Y, Lee SM, Park M, Choi HJ, Kang S, Choi BI, Lew H. Treatment of traumatic optic neuropathy using human placenta-derived mesenchymal stem cells in Asian patients. Regen Med. 2020 Oct;15(10):2163-2179. doi: 10.2217/rme-2020-0044. Epub 2020 Dec 14. PMID 33315474
- [Background] Zhao T, Liang Q, Meng X, Duan P, Wang F, Li S, Liu Y, Yin ZQ. Intravenous Infusion of Umbilical Cord Mesenchymal Stem Cells Maintains and Partially Improves Visual Function in Patients with Advanced Retinitis Pigmentosa. Stem Cells Dev. 2020 Aug;29(16):1029-1037. doi: 10.1089/scd.2020.0037. Epub 2020 Jul 15. PMID 32679004
- [Background] Ozmert E, Arslan U. Management of retinitis pigmentosa by Wharton's jelly derived mesenchymal stem cells: preliminary clinical results. Stem Cell Res Ther. 2020 Jan 13;11(1):25. doi: 10.1186/s13287-020-1549-6. PMID 31931872